CLINICAL TRIAL: NCT02338791
Title: Rehabilitative Ultrasound Imaging: Measurements of Articular Movement of the Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Dexter Witt, Associate Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-1211
Record Dates: First submitted 2015-01-05; First posted 2015-01-14 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Disorder of Shoulder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Manual Mobilization (Experimental): Grade I, II and III manual mobilizations in the inferior, posterior and distractive directions.
  Interventions: Device: Manual Mobilization

INTERVENTIONS:
Device: Manual Mobilization — Stabilization of the glenoid fossa with movement of the humerus using varying degrees of force as applied by a physical therapist. Subject is positioned with the shoulder in 55 degrees of abduction and 30 degrees of horizontal adduction. Manual force is applied by a physical therapist on the proximal humeral head moving the humeral head posterior, inferior or lateral (distraction). An ultrasound transducer placed over the anterior shoulder joint provides imaging of the humeral head and the glenoid fossa. This manual intervention is repeated three times in each direction on each arm.

SUMMARY:
The purpose of this study is to measure the amount of movement between the bones of the shoulder joint when mobilization techniques are applied by a physical therapist.

DETAILED DESCRIPTION:
The purpose of this study is to image the articular joint movement of the glenohumeral joint utilizing ultrasound imaging (USI). Specific aims include: 1) measurement of the distance between the articular surfaces at rest; 2) measurement of the distance between the articular surfaces during manually applied glides of those surfaces; and 3) analysis of any association between the amount of glide and reported joint mobility, force application, or joint position.

Subjects will be recruited from a population of convenience. After consenting to participate, eligible subjects will complete a demographic questionnaire and pretesting of scapular and shoulder mobility. Two days of testing will be scheduled. On the first day, three grades of glenohumeral mobilization will be applied in the following directions: distraction, posterior and inferior. A handheld dynamometer will measure force; ultrasound imaging will record glenohumeral joint position. Each grade and direction will be repeated three times on the right and the left shoulder. On the second day, the mobilizations will be repeated. Measurements of humeral movement will be calculated from the ultrasound images.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic subjects with no history of neck, shoulder, or arm pain; full active pain free range of motion at the cervical spine and shoulders

Exclusion Criteria:

* neuromuscular or musculoskeletal disorders; connective tissue disorders such as rheumatoid arthritis; inflammatory conditions such as Crohns disease; Down's syndrome; Marfan's syndrome; medically diagnosed hypermobility; history of neck, shoulder or arm trauma, pain, or surgery including dislocation and rotator cuff tears; pregnancy; and metal implants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Movement of the humeral head | Immediate measurement of humeral head movement concurrent with application of manual mobilization
  The movement of the humeral head in reference to the glenoid fossa is recorded using ultrasound imaging. The amount of movement (as measured in millimeters) between the image taken on rest and the image taken during the manual mobilization is calculated for each direction of manual mobilization. This primary outcome measure is obtained during the performance of the manual mobilization. Subjects are tested and this primary outcome measured during the intervention (manual mobilization) on Day one and, within one week, on Day two. Each subject participates in the study for approximately one week.

SECONDARY OUTCOMES:
Force of Mobilization | Immediate measurement of force used during the application of manual mobilization
  Amount of force used during the application of grade I, grade II and grade III mobilizations. The maximal force used during the performance of the manual mobilization (as measured in Newtons) is recorded using a hand held dynamometer as the mobilization is performed. Subjects are tested and this secondary outcome measured during the intervention (manual mobilization) on Day one and, within one week, on Day two. Each subject participates in the study for approximately one week.

CONTACTS AND LOCATIONS:
Overall Officials: Dexter Witt, DHS, Principal Investigator — University of Cincinnati; Nancy Talbott, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No